CLINICAL TRIAL: NCT05692336
Title: a Comparison Between the Effectiveness of Vestibular Versus Dual Task Training on Balance in Children With Diplegic Cerebral Palsy
Brief Title: a Comparison Between the Effectiveness of Vestibular and Dual Task on Balance in Diplegic Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amira Ashraf Mahmoud Mohamed, teaching assisstant at faculty of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/003716
Record Dates: First submitted 2022-12-22; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Diplegic Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vestibular training (Experimental): balance training that focus on vestibular system stimulation like when the eyes are folded while standing on a balance board or walking on swinging boards
  Interventions: Other: vestibular training
- dual task training (Experimental): The children received special balance training in the form of dual-task training performing balance activities as a basic task in conjunction with second task that includes upper limb activity using basketball and long rings shaft or cognitive task like telling a story during balance training .
  Interventions: Other: dual task training

INTERVENTIONS:
Other: vestibular training — balance training in the form of vestibular training
  Arms: vestibular training
Other: dual task training — balance training in the form of dual task training
  Arms: dual task training

SUMMARY:
the study is carried out to identify If there is any difference between the effectiveness of Vestibular training and Dual task training on balance in children with Diplegic Cerebral Palsy.

so in this study the sample will be divided into two equal groups, each group will recieve only one type of training ( vestibular training or dual task training ) the balance of the diplegic children will be assessed before and after using HUMAC balance system and pediatric balance scale , the results will be compared between both groups and if there is one training is more effective than the other , it will be recommended most in the future treatment program.

DETAILED DESCRIPTION:
A comparative experimental design was used. Children participating in this study were assigned into two equal groups, Thirty four children with diplegic Cerebral Palsy of both genders who have balance problems were selected to join this study with the following criteria:

1. all the children diagnosed as diplegic cerebral palsy.
2. Their age are range from 5 to 10 years old.
3. The degree of spasticity is between grade 1 or 1+ according to Modified Ashworth Scale (Charalambous ,2013).
4. They are at level I OR II on Gross Motor Function Classification System .
5. All the children were able to follow verbal command and instructions.

And Children were excluded in the presence of the following:

1. Children that suffer from epilepsy.
2. Severe visual and auditory problems.
3. Structural or fixed soft tissue deformities of Lower extremities.
4. Severe mental retardation.
5. Botox injection in the lower extremity in the past 6 months..

all the children will be assigned in one of two groups ( vestibular training group and dual task group ) the training will be continue for definite period of time , and the balance abilities for the children in each group will be assessed before and after the treatment completely ended and the result will be compared to conclude which group benefit more and have a greater balance improvement and the treatment that causes a greater improvement will be more recommended in the future physical therapy plan for treatment of diplegic cerebral palsied children.

the balance is assessed using HUMAC balance system and pediatric balance scale .

ELIGIBILITY:
Inclusion Criteria:

1. clinical diagnosis of diplegic cerebral palsy .
2. age range : from 5 to 10 years old.
3. The degree of spasticity is between grade 1 or 1+ according to Modified Ashworth Scale (Charalambous ,2013).
4. They are at level I OR II on Gross Motor Function Classification System .
5. All the children were able to follow verbal command and instructions.

Exclusion Criteria:

1. Children that suffer from epilepsy.
2. Severe visual and auditory problems.
3. Structural or fixed soft tissue deformities of Lower extremities.
4. Severe mental retardation.
5. Botox injection in the lower extremity in the past 6 months

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Estimated)
Dates: Start 2022-02-20 (Actual); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Static Balance | 2 months of training
  static balance will be assessed using HUMAC balance system , a comparison of the results between two groups will be carried out , and the more effective treatment program will be more recommended than the other
dynamic balance | 2 months of training
  dynamic balance will be assessed using pediatric balance scale and a comparison between the results of the two groups will be done to recommend one over the other.
which training will be more beneficial for the diplegic child balance | 2 months
  after the results of both groups (for static and dynamic balance) are analyzed one treatment will be recommended most (the treatment for the group that has greater balance improvement ).

CONTACTS AND LOCATIONS:
Overall Officials: amira A mahmoud, Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical Therapy Cairo University, Giza, Egypt